CLINICAL TRIAL: NCT06373640
Title: HAPTO Study: Haemoglobin And Vancomycin Pharmacokinetics in the Cerebrospinal Fluid Following Subarachnoid Haemorrhage: Therapeutic Optimisation of Haptoglobin
Brief Title: Haemoglobin And Vancomycin Pharmacokinetics in the Cerebrospinal Fluid Following Subarachnoid Haemorrhage
Acronym: HAPTO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RHM NEU0458
Record Dates: First submitted 2024-04-16; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Subarachnoid Hemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EVD first (Other): Vancomycin to be administered first through an EVD
  Interventions: Procedure: Insertion of drains; Drug: Vancomycin
- Lumbar drain first (Other): Vancomycin to be administered first through a lumbar drain
  Interventions: Procedure: Insertion of drains; Drug: Vancomycin

INTERVENTIONS:
Procedure: Insertion of drains — Insertion of lumbar drain and basal cistern drain
  Other Names: Drain insertion
Drug: Vancomycin — Administration of vancomycin
  Other Names: Antibiotic adminsitration

SUMMARY:
The HAPTO study will recruit adult patients with aSAH due to a burst aneurysm. These patients must be scheduled to have their aneurysm treated surgically to prevent further bleeds, and need an external ventricular drain for clinical reasons (to drain fluid and relieve pressure on the brain). At the end of their surgery for their aneurysm, a further drain will be left at the site of the surgery (which is in the basal cisterns) and they will additionally have a drain sited in their lumbar spine. Vancomycin will be given through these drains. Additionally, these drains will allow the fluid in the brain to be collected to measure how haemoglobin levels and vancomycin levels differ between compartments and change over time. Patients will participate in the study over a period from recruitment at three days after aSAH to a maximum of ten days after aSAH. The data will be analysed to determine the relationship in haemoglobin concentrations between different areas of the brain and spine after aSAH, and how vancomycin distribution is related to its route of administration.

DETAILED DESCRIPTION:
The HAPTO study aims to improve the treatment of a specific type of stroke known as aneurysmal subarachnoid haemorrhage (aSAH). This stroke can occur when a weak point in a blood vessel in the brain called an aneurysm bursts. This causes bleeding into the surrounding area. aSAH is not only life-threatening, but also leaves many survivors with long-term disabilities and health issues that affect the quality of their life.

After aSAH, haemoglobin - a protein normally found inside red blood cells - leaks out into the brain and its surrounding fluid. While inside red blood cells, haemoglobin is safe, but when it leaks out it is toxic and causes more damage to the brain. Our bodies have a natural defence, which is a substance called haptoglobin. Haptoglobin can grab onto haemoglobin and potentially stop its harmful effects. Although there is lots of haptoglobin in the rest of the body, there is virtually none in the brain to protect against haemoglobin. Therefore, haptoglobin is being developed as a drug that can be delivered directly to the brain to treat patients with aSAH.

The HAPTO study measures the amount of haemoglobin that different areas of the brain and spine are exposed to after aSAH. These areas are the ventricles (cavities in the brain), the lumbar spine (lower back), and the basal cisterns (near the brain's base where aneurysms are normally found). By collecting fluid samples from these places, we can measure how much haemoglobin there is, and from this, we can work out how much haptoglobin will be needed.

Apart from knowing how much to give, we need to know where to give it. The main options are to insert it either through a tube in the cavities of the brain (external ventricular drain) or a tube inserted into the spine (lumbar drain). Little is known about how drugs distribute around the nervous system in general, and even less in patients who have had an aSAH in whom the flow of fluid around the brain is disturbed. This study will try to find out more by using a common antibiotic, vancomycin, as a tracer to understand how drugs move within different regions of the brain and spine following aSAH. This approach will provide valuable insights into the possible ways to give haptoglobin (and any other future treatments requiring injection into the brain or spine).

The HAPTO study will recruit adult patients with aSAH due to a burst aneurysm. These patients must be scheduled to have their aneurysm treated surgically to prevent further bleeds, and need an external ventricular drain for clinical reasons (to drain fluid and relieve pressure on the brain). At the end of their surgery for their aneurysm, a further drain will be left at the site of the surgery (which is in the basal cisterns) and they will additionally have a drain sited in their lumbar spine. Vancomycin will be given through these drains. Additionally, these drains will allow the fluid in the brain to be collected to measure how haemoglobin levels and vancomycin levels differ between compartments and change over time. Patients will participate in the study over a period from recruitment at three days after aSAH to a maximum of ten days after aSAH. The data will be analysed to determine the relationship in haemoglobin concentrations between different areas of the brain and spine after aSAH, and how vancomycin distribution is related to its route of administration.

ELIGIBILITY:
Inclusion Criteria:

* aSAH on pre-repair CT scan graded 2, 3, or 4 on Modified Fisher Scale (diffuse [clot present in both hemispheres] thick or thin, or local thick).
* Ruptured saccular aneurysm confirmed by angiography (CT angiogram, MR angiogram, or digital subtraction angiography)
* EVD in situ in the lateral ventricle (or anticipated to have an EVD inserted)
* Scheduled for surgery to clip the aneurysm (or has had surgery to clip the aneurysm with a proximal Sylvian fissure/basal cistern drain left in situ)
* CT scan completed after aneurysm repair to confirm EVD position and exclude major post-repair complications
* Aged 18 years to 80 years (inclusive) at the time of providing written informed consent.
* Capable of providing written (or electronic) informed consent and willing and able to adhere to all protocol requirements or informed consent provided by the subject's legally authorized representative if the subject lacks capacity at the time of screening.
* Haemodynamically stable after resuscitation, with systolic blood pressure ≥ 90 mm Hg at screening

Exclusion Criteria:

* SAH due to giant aneurysm (i.e., size ≥ 2.5 cm) or causes other than a saccular aneurysm (e.g., rupture of infective aneurysm, traumatic head injury / traumatic SAH).
* Bilateral blown pupils
* Isolated intraventricular haemorrhage or intracerebral haemorrhage without SAH
* aSAH diagnosed on LP with no evidence of blood on CT
* Bleeding disorder
* Decompressive hemicraniectomy at screening
* Contraindications to vancomycin: known hypersensitivity to vancomycin or teicoplanin, documented history of hearing impairment, wearing a hearing aid, or renal insufficiency (estimated glomerular filtration rate <60 ml/min/1.73m2)
* Pregnant, planning to become pregnant, or breastfeeding
* Underwent prophylactic hypertension or balloon angioplasty between admission to hospital for aSAH and screening
* Given therapeutic magnesium infusion, and other intrathecal or intraventricular vasodilators or thrombolytics between admission to hospital for aSAH and screening
* Given IV or intrathecal / intraventricular nicardipine between admission to hospital for aSAH and screening
* Given antifibrinolytics (e.g., tranexamic acid) or intrathecal thrombolytics between admission to hospital for aSAH and screening
* Current participation in an interventional clinical study
* Direct involvement in the planning and / or conduct of this study (e.g., Sponsor employees, study site staff, as well as their immediate family members [i.e., spouse, parent, child, or sibling, whether biological or legally adopted]).
* Any medical condition or other issue that, in the opinion of the Investigator and / or Sponsor, would render the subject unsuitable for participation in the study (ie, issue may compromise subject safety or compliance, impede study conduct, or interfere with interpretation of study results).
* Subject met eligibility criteria but was not needed for enrolment / randomization.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
CSF-haemoglobin concentration | 3 days to 10 days
  CSF-haemoglobin concentration

IPD SHARING:
Plan to Share IPD: No